CLINICAL TRIAL: NCT06270290
Title: Observational Cross-sectional Study Investigating the History of Concussion and Exposure to Contact Sports in Patients With REM Sleep Behaviour Disorder (RBD) Versus Controls (Without a Diagnosis of RBD)
Brief Title: The COSP-RBD Study: Concussions and Contact Sports in RBD vs Controls
Acronym: COSP-RBD
Status: Recruiting | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 327648
Record Dates: First submitted 2024-02-13; First posted 2024-02-21 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: REM Sleep Behavior Disorder; Concussion, Brain
Keywords: REM sleep behaviour disorder; concussion; contact sports
MeSH Terms: conditions — REM Sleep Behavior Disorder; Brain Concussion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RBD group: Participants with a diagnosis of REM sleep behaviour disorder
  Interventions: Other: Exposure to contact sports or history of concussions
- Control group: Participants without a diagnosis of REM sleep behaviour disorder
  Interventions: Other: Exposure to contact sports or history of concussions

INTERVENTIONS:
Other: Exposure to contact sports or history of concussions — History of contact sports practices or of concussions

SUMMARY:
The goal of this observational study is to investigate concussions and contact sports practices in REM sleep behaviour disorder (RBD).

The main questions it aims to answer are:

* What is the proportion of patients with RBD that have a history of concussions or exposure to contact sports?
* Is this proportion higher to that in control patients without a diagnosis of RBD?

Participants will undergo an interview with a sleep medicine specialist to answer questions about history of concussions and contact sports practices.

Researchers will compare an RBD group and a control group (without RBD) to see if the proportion of concussions and exposure to contact sports differ.

DETAILED DESCRIPTION:
Rapid eye movement (REM) sleep behaviour disorder (RBD) is a parasomnia characterised by the presence of acting-out behaviours in sleep and vivid dreams, which diagnosis requires the demonstration of loss of REM atonia or an RBD episode on a video-polysomnography (v-PSG). Importantly, patients with the isolated form of RBD are at a high risk to develop Parkinson's disease or related neurodegenerative conditions, such as dementia with Lewy bodies or multiple system atrophy (synucleinopathies). Hence, RBD is a condition frequently associated to, and often preceding, a manifest neurodegenerative disorder. It is therefore extremely relevant to identify factors that may be linked to these early neuropathological processes. This will be key for a timely diagnosis of isolated RBD, especially when neuroprotective trials become available.

There is also solid evidence showing that repeated concussions lead to an increased risk to develop a neurodegenerative disorder such as Parkinson's disease, chronic traumatic encephalopathy, all-causes of dementia, and amyotrophic lateral sclerosis.

In epidemiological studies, self-reported head injury was more frequently present in RBD vs controls. Head injury was also proposed as a possible risk factor for probable RBD in large community-based studies, although the diagnosis of RBD was not confirmed by v-PSG in these cases. Of note, a higher frequency of professional football players was demonstrated on a recent study including a large cohort of RBD patients when compared to a control group. Moreover, in a group of deceased contact sport athletes with neuropathology diagnosing traumatic chronic encephalopathy, probable RBD was present in over 30% of the sample.

We hypothesise that the presence of a history of concussions or exposure to contact sports is more frequently reported by patients with v-PSG-confirmed RBD than by sex- and age-matched controls. There is, however, a lack of further characterisation of the head-impact events and circumstances in which they have occurred. It would be relevant to know whether repeated head impacts while playing contact sports or concussions that may have not been formally diagnosed, and that may have happened in non-professional as well as in professional sport activities, may be linked with RBD. The demonstration of a higher percentage of concussions or exposure to contact sports in RBD would provide greater evidence related to neuropathological changes in the context of certain sport practices.

Given the prognostic implications of a diagnosis of RBD and the established links between head injury and neurodegenerative conditions, it seems relevant to assess the characteristics of previous concussions or exposure to head-impact sports in patients with v-PSG-confirmed RBD. This will provide further evidence to help increase the awareness of RBD (hopefully leading to a more timely diagnosis of this condition), and potentially aid the development of health and government policies, including those relating to safer sport practices.

As one of the major sleep disorders centres in the UK, and one of the few with expertise in sleep neurological conditions such as RBD, it is our responsibility to assess and report our experience on this matter.

The primary objective of this study is to assess the frequency of self-reported history of concussions or exposure to contact sports in patients with v-PSG-confirmed RBD against a control group (without a diagnosis of RBD).

Secondary objectives of this study will include investigating concussions/head impact characteristics in RBD vs control group. We will also aim to search differences in demographic and clinical variables between RBD patients with and without history of concussions/head impact.

ELIGIBILITY:
Inclusion criteria group with RBD:

* Patient at the SDC with diagnosis of RBD (Guy's and St Thomas' NHS Foundation Trust).
* 50 years of age or above (patients below this age would not be expected to have a RBD related to a synucleinopathy and other causes of RBD would need to be considered instead - e.g. narcolepsy, post-traumatic stress disorder).

Inclusion criteria control group:

* Patients who have undergone a v-PSG at the SDC (Guy's and St Thomas' NHS Foundation Trust) and who do not have history of suspected RBD or RBD confirmed by v-PSG.
* 50 years of age or above This group will be age- and sex-matched to the RBD group.

Exclusion criteria group with RBD:

* Age < 50 years of age.
* Diagnoses of narcolepsy or post-traumatic stress disorder.
* Subjects lacking capacity or literacy.
* Non-English speakers.

Exclusion criteria control group:

* Age < 50 years of age (in order to match RBD group).
* REM sleep without atonia or confirmed RBD on v-PSG.
* Diagnosis of neurological diseases, cognitive complaints or motor complaints.
* Clinical history suggestive of parasomnia that may be included in the differential of RBD.
* Subjects lacking capacity or literacy.
* Non-English speakers.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of RBD at the Sleep Disorders Centre (Guy's and St Thomas' NHS Foundation Trust) will be identified via the sleep clinics. Expected number of eligible participants are 100, from which we expect 80 to agree to participate.
  An age- and sex-matched control group of 60 participants will be obtained also via the Sleep Disorders Centre clinics (Guy's and St Thomas' NHS Foundation Trust).
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2024-04-23 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of history of contact sports practice / concussion in RBD and control participants. | 1 year
  Proportion of self-reported history of concussions or exposure to contact sports in participants with v-PSG-confirmed RBD and that in a control group (without a diagnosis of RBD).

SECONDARY OUTCOMES:
Differences in concussions characteristics between RBD and control participants. | 1 year
  Concussions/head impact characteristics differences (as per interview designed for this study) in RBD and control participants.
Demographic or clinical differences between RBD participants with and without concussions history. | 1 year
  Demographic and clinical differences between RBD participants with and without history of concussions/head impact: age, sex, age at RBD onset and diagnosis, cardiovascular comorbidities, antidepressant or betablocker use at RBD onset, smoking status, alcohol intake, history of recreational substance misuse, history of sport-related supplements or substances use, education level, family history of neurodegenerative conditions, diagnosis of established neurodegenerative condition, time since diagnosis of RBD to neurodegenerative condition.

CONTACTS AND LOCATIONS:
Overall Officials: Gillian Radcliffe, Study Chair — Guys and St. Thomas NHS Foundation Hospital
Locations (1):
- Guy's & St Thomas' NHS Foundation Trust, London, United Kingdom